CLINICAL TRIAL: NCT04937205
Title: Understanding Motivation for Exercise to Enhance Physical Activity Adherence in Adults With Obesity
Brief Title: Motivation for Exercise and Physical Activity Adherence
Acronym: MOVE
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19-0826; F32DK122652 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Obesity
Keywords: Physical activity; Motivation; Exercise
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 2: This group of study participants started the 52-week parent randomized controlled trial (NCT03411356) on February 13, 2019.
  Interventions: Behavioral: MOVE
- Cohort 3: This group of study participants started the 52-week parent randomized controlled trial (NCT03411356) on November 5, 2019.
  Interventions: Behavioral: MOVE
- Cohort 4: This group of study participants started the 52-week parent randomized controlled trial (NCT03411356) on October 22, 2020.
  Interventions: Behavioral: MOVE

INTERVENTIONS:
Behavioral: MOVE — The MOVE physical activity support program is based on the Self-Determination Theory and targets autonomous motivation for physical activity by encouraging 1) choice in physical activity type (e.g. walking, household chores, yoga), 2) a meaningful, value-based rationale for engaging in physical activity, and 3) physical activity that is intrinsically enjoyable. MOVE was delivered during two, 60-75 minute group-based classes and one, 45 minute individualized 1:1 support session to enhance adherence to physical activity recommendations within a lifestyle weight loss program. The group-based classes included a combination of PowerPoint slides, participant handouts, and group-based discussions. All MOVE content was delivered by trained study staff.

SUMMARY:
The limited success of our current approaches to increase adoption and maintenance of physical activity in adults with overweight and obesity is a substantial barrier to effectively address the current obesity epidemic. This mentored F32 application addresses the significant public health issue of obesity and associated risk of major chronic diseases by using mixed methods research to optimize an innovative, theoretically based physical activity intervention designed to enhance motivation for exercise in adults with overweight and obesity.

DETAILED DESCRIPTION:
Physical activity (PA) is one of the best predictors of sustained weight loss and current guidelines recommend high levels of PA to prevent weight regain after weight loss. However, long-term adherence to PA is generally poor when adults with overweight/obesity are provided an exercise prescription consistent with current guidelines. Thus, it is essential to evaluate novel strategies to enhance adoption and maintenance of PA in adults with overweight/obesity. The overall goal of this mentored F32 application is to use mixed methods research to optimize an innovative, theoretically based PA intervention designed to enhance motivation for exercise in adults with overweight/obesity. Specifically, the objectives of this proposal are to evaluate and optimize a theory-based PA intervention (called MOVE) designed to enhance motivation for exercise as a sub-study of an ongoing weight loss "parent" trial (COMIRB, Protocol #17-0369). In Aim 1, adults from an ongoing behavioral weight loss trial (R01DK111622) will receive the MOVE intervention and participate in focus groups to explore how participants experience MOVE. In Aim 2, we will use a mixed methods convergent design to integrate quantitative results from a secondary data analysis and qualitative results (Aim 1) to optimize MOVE in preparation for a full evaluation of MOVE in a future randomized controlled study.

ELIGIBILITY:
Inclusion Criteria:

* A current study participant randomized to the parent trial in cohorts 2-4 for COMIRB, Protocol #17-0369
* Completed at least 2 of 3 MOVE program components (attended ≥80% of either group-based class and/or attended the one-on-one support session).

Exclusion Criteria:

* None

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Volunteers from the parent trial who are eligible and willing to participate were included in the focus groups. To achieve aim 1 of this proposal, participants randomized to cohorts 2-4 of the parent study who have completed at least 2 of the 3 MOVE components were invited to participate in a focus group.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2021-04-14 (Actual); Study Completion 2021-04-14 (Actual)

PRIMARY OUTCOMES:
Acceptability | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about their satisfaction with major aspects of the MOVE physical activity support program including: 1) MOVE content and 2) delivery of MOVE content including meeting frequency and structure for both group-based and 1:1 meetings. Participants were also asked about their overall experience with the MOVE program, things that worked well, things that did not work well, and about the most important things they learned from the MOVE program.

SECONDARY OUTCOMES:
Motivation for Physical Activity | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about reasons why they want to be physically activity.
Motivation for Sedentary Behavior | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about reasons why they want to be sedentary.
Barriers to Physical Activity | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about things that make it harder for them to add more physical activity into their daily lives.
Facilitators to Physical Activity | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about things that make it easier for them to add more physical activity into their daily lives.
Perceptions of Physical Activity Messages | weeks 21-30
  During a 90-minute semi-structured focus group, participants were asked about their perception of two different physical activity messages:
  1. "For substantial health benefits, adults should do at least 150 minutes (2 hours and 30 minutes) to 300 minutes (5 hours) a week of moderate-intensity, or 75 minutes (1 hour and 15 minutes) to 150 minutes (2 hours and 30 minutes) a week of vigorous-intensity aerobic physical activity, or an equivalent combination of moderate- and vigorous-intensity aerobic activity. Preferably, aerobic activity should be spread throughout the week."
  2. "Move in ways that make you feel good. Benefits of physical activity include improved mood, sleep, less anxiety, more patience. All movement counts. Find opportunities to move throughout the day."
Influence of Diet on Physical Activity Adherence | weeks 21-30
  Participants were asked about how their randomization to their diet strategy (either intermittent fasting or daily caloric restriction) impacted their ability to adhere (or not adhere) to physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Danielle M Ostendorf, PhD, Principal Investigator — University of Colorado Anschutz Health and Wellness Center
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No